CLINICAL TRIAL: NCT03639090
Title: Mass Spectrometry Detection of Drugs in Single Bladder Cancer Cells From Patients
Brief Title: Mass Spectrometry in Single Bladder Cancer Cells
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Mass Spectrometry; 1R21CA204706-01 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-08-20 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Bladder Cancer
Keywords: chemotherapy, mass spectrometry
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine sample, blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: mass spectrometry — mass spectrometry for bladder cancer cells

SUMMARY:
The study is a pilot study in the feasibility of a diagnostic technique. There is no current data on detection of cisplatin in cancer cells derived from human urine. This study will generate preliminary data so that future studies may be done with more definitive end points in mind.

DETAILED DESCRIPTION:
The aim of this study is to determine the feasibility of using a novel mass spectrometry instrument to measure the intracellular concentration of chemotherapeutic drug within an active tumor cell. If successful, this technique could be applied to dosage streamlining in patients and customization of dosage based on individual tumor characteristics. It also opens the door to research on novel chemotherapy agents or agents not typically used in a specific malignancy to determine if therapeutic levels can be obtained in tumor cells.

Personalized chemotherapy is an evolving field with the underlying goal being minimization of side effects of treatment while maximizing net patient benefit for therapy. A key difficulty in personalized chemotherapy is that the determination of therapeutic benefit comes well after the administration of treatment has been completed. For most forms of chemotherapy there does not exist a laboratory study that can determine the concentration of therapeutic agent within the tumor itself and as such, real time dose adjustments are based only on toxicity, not on tumor penetrance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of bladder cancer
2. Patients must be undergoing their first cycle of cisplatin based chemotherapy due to metastatic disease or as pre-operative treatment before cystectomy
3. Patients with a diagnosis of bladder cancer who will not be undergoing chemotherapy
4. Patients must have demonstrated positive urinary cytology prior to inclusion in the study

Exclusion Criteria:

1. Patients who do not have bladder cancer.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bladder cancer at Stephenson Cancer who are undergoing treatment with cisplatin are eligible to participate.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the intracellular concentration | 4 years
  An instrument to determine the concentration of therapeutic agent will be used. Results of the test will be used to determine feasibility of this technique for application in personalized chemotherapy dosing and treatment monitoring in the future. For each patient sample, the concentration of cisplatin will be measured in several different cells, as many as 10 depending upon the characteristics of the sample. The results of each individual run of the test will be recorded for the purpose of verifying internal consistency of the technique. Measurement will be first in relative mass of the agent to other known controls which will be used to calculate the approximate cellular concentration of cisplatin. Refining the technique for estimating the concentration is one of the goals of the project.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Heinlen, M.D., Principal Investigator — University of Oklahoma HSC, Department of Urology
Locations (1):
- University of Oklahoma HSC, Department of Urology, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No